CLINICAL TRIAL: NCT03741829
Title: TS Overexpression in SCLC: Mechanism and Therapeutic Targeting
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00043264; Pilot Funds 11347 (Other Grant/Funding Number: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH); CCCWFU 62A17 (Other: NCI)
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Thymidylate Synthase; Cancer; Cancer Treatments
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be extracted from the PDX tumor and from the blood sample obtained from the same subject/patient. Both samples will undergo DNA sequencing in the Cancer Genomics Shared Resource. The DNA sequences will be compared to differentiate between tumor-specific mutations and germ-line polymorphisms from the same individual. The mutation profile is characteristic of the tumor and will also be used to test for genetic drift as the PDX tumor is propagated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Samples from transbronchial Biopsy: Samples from participants with SCLC.

SUMMARY:
The purpose of this research study is to determine the amount of a protein named thymidine synthase that is being made by cancer and to develop laboratory models called PDX (patient derived xenografts) to learn more about SCLC (small cell lung cancer) and to begin testing new treatments.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is a highly lethal malignancy that is not treatable with targeted therapies and that does not respond long-term to treatment with cytotoxic chemotherapy1. One distinguishing molecular characteristic of SCLC is very high expression levels of thymidylate synthase (TS). TS plays an important role in de novo nucleotide biosynthesis and the very high TS levels expressed in SCLC cells indicate that these cells require the de novo nucleotide biosynthetic pathway to proliferate. Thus, complete TS inhibition could result in highly favorable outcomes in SCLC patients. TS inhibitors have been evaluated in SCLC clinical trials and have anti-tumoral activity when combined with a second chemotherapeutic agent. However, treatment with TS inhibitors has not been shown to surpass other combination chemotherapy regimens. An important point regarding these clinical studies is that TS activity levels were not monitored as an endpoint of drug response, thus it is not known whether TS activity was efficiently inhibited.Investigators predict that complete TS inhibition will result in favorable outcomes.

With support from Wake Innovations, Investigators are developing a novel fluoropyrimidine polymer, CF10, which strongly inhibits TS. CF10 is a second generation fluoropyrimidine polymer. The first generation polymer, F10, showed excellent anti-cancer activity in animal models of acute myeloid leukemia, glioblastoma, and prostate cancer. CF10 is designed to have improved tumor penetration and better in vivo stability than F10. Investigators hypothesize that CF10 will be highly effective for treating SCLC both as a single agent and in combination with TS inhibitors that target alternative sites of the TS enzyme.

After establishing CF10 has activity as a single agent and in combination with folate-based TS inhibitors (e.g. pemetrexed) in SCLC cell lines and xenograft models, Investigators will test CF10 in patient-derived xenograft (PDX) models and in organoids derived from SCLC patient samples. Investigators will develop PDX models of SCLC and SCLC organoids using transbronchial fine needle aspiration (FNA) from SCLC patients at Baptist/WFBCCC collected by co-I's Bellinger, Dotson, and Thomas. Non-malignant cells will be collected using a brush biopsy to enable comparison of malignant and non-malignant tissue from the same patient with regard to mechanistic endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a diagnostic FNA by the following diagnostic modalities utilizing FNA: Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS- TBNA) or conventional transbronchial FNA.
* Patients must have radiographic evidence for presumed lung cancer or have a previously diagnosed SCLC with clinical evidence of recurrence. Patients undergoing FNA of potential SCLC metastates to lymph nodes are also included (e.g., patients with abnormal mediastinal lymphadenopathy). FNA biopsies from separate locations in the same patient will be considered separate specimens.
* Age >18 years. Used to define adult age that can independently provide consent.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients whose FNA biopsy is unable to provide classification by pathology or is non-diagnostic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Women and men of all races and ethnicity who meet the above-described eligibility criteria are eligible for this trial.
  * The study consent form will also be provided in Spanish for Spanish-speaking participants.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-01-03 (Actual)

PRIMARY OUTCOMES:
TYMS (Thymidylate Synthetase) expression levels | After biopsy collection, up to 1 year
  TYMS (Thymidylate Synthetase) expression levels will be measured on biopsied malignant tissue as well as non-malignant tissue.
miRNA expression levels | After biopsy collection, up to 1 year
  miRNA expression levels will be measured on biopsied malignant tissue as well as non-malignant tissue.

OTHER OUTCOMES:
Survival of mice at 60 days implanted with tumor and treated with CF10 | 60 days
Number of samples with PDX model development | After biopsy collection, up to 1 year
Levels of TS activity | After biopsy collection, up to 1 year
Levels of Top1cc | After biopsy collection, up to 1 year
Levels of DNA double strand breaks | After biopsy collection, up to 1 year
Tumor volume | After biopsy collection, up to 1 year
Number of apoptotic cells. | After biopsy collection, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: William Gmeiner, Ph.D, MBA, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asai N, Ohkuni Y, Kaneko N, Yamaguchi E, Kubo A. Relapsed small cell lung cancer: treatment options and latest developments. Ther Adv Med Oncol. 2014 Mar;6(2):69-82. doi: 10.1177/1758834013517413. PMID 24587832
- [Background] Byers LA, Wang J, Nilsson MB, Fujimoto J, Saintigny P, Yordy J, Giri U, Peyton M, Fan YH, Diao L, Masrorpour F, Shen L, Liu W, Duchemann B, Tumula P, Bhardwaj V, Welsh J, Weber S, Glisson BS, Kalhor N, Wistuba II, Girard L, Lippman SM, Mills GB, Coombes KR, Weinstein JN, Minna JD, Heymach JV. Proteomic profiling identifies dysregulated pathways in small cell lung cancer and novel therapeutic targets including PARP1. Cancer Discov. 2012 Sep;2(9):798-811. doi: 10.1158/2159-8290.CD-12-0112. Epub 2012 Sep 6. PMID 22961666
- [Background] Tanaka F, Wada H, Fukui Y, Fukushima M. Thymidylate synthase (TS) gene expression in primary lung cancer patients: a large-scale study in Japanese population. Ann Oncol. 2011 Aug;22(8):1791-7. doi: 10.1093/annonc/mdq730. Epub 2011 Feb 14. PMID 21321092
- [Background] Socinski MA, Weissman C, Hart LL, Beck JT, Choksi JK, Hanson JP, Prager D, Monberg MJ, Ye Z, Obasaju CK. Randomized phase II trial of pemetrexed combined with either cisplatin or carboplatin in untreated extensive-stage small-cell lung cancer. J Clin Oncol. 2006 Oct 20;24(30):4840-7. doi: 10.1200/JCO.2006.07.7016. PMID 17050869
- [Background] Pardee TS, Gomes E, Jennings-Gee J, Caudell D, Gmeiner WH. Unique dual targeting of thymidylate synthase and topoisomerase1 by FdUMP[10] results in high efficacy against AML and low toxicity. Blood. 2012 Apr 12;119(15):3561-70. doi: 10.1182/blood-2011-06-362442. Epub 2012 Feb 23. PMID 22362039
- [Background] Gmeiner WH, Debinski W, Milligan C, Caudell D, Pardee TS. The applications of the novel polymeric fluoropyrimidine F10 in cancer treatment: current evidence. Future Oncol. 2016 Sep;12(17):2009-20. doi: 10.2217/fon-2016-0091. Epub 2016 Jun 9. PMID 27279153
- [Background] Gmeiner WH, Lema-Tome C, Gibo D, Jennings-Gee J, Milligan C, Debinski W. Selective anti-tumor activity of the novel fluoropyrimidine polymer F10 towards G48a orthotopic GBM tumors. J Neurooncol. 2014 Feb;116(3):447-54. doi: 10.1007/s11060-013-1321-1. Epub 2013 Dec 18. PMID 24346635
- [Background] Gmeiner WH, Willingham MC, Bourland JD, Hatcher HC, Smith TL, D'Agostino RB Jr, Blackstock W. F10 Inhibits Growth of PC3 Xenografts and Enhances the Effects of Radiation Therapy. J Clin Oncol Res. 2014 Jul-Aug;2(4):1028. PMID 26020060
- [Background] Anderson WC, Boyd MB, Aguilar J, Pickell B, Laysang A, Pysz MA, Bheddah S, Ramoth J, Slingerland BC, Dylla SJ, Rubio ER. Initiation and characterization of small cell lung cancer patient-derived xenografts from ultrasound-guided transbronchial needle aspirates. PLoS One. 2015 May 8;10(5):e0125255. doi: 10.1371/journal.pone.0125255. eCollection 2015. PMID 25955027